CLINICAL TRIAL: NCT01595217
Title: The Incremental Value of 3T Diffusion-Weighted MRI in Diagnosing Extrahepatic Cholangiocarcinoma
Brief Title: MRCP Diagnoses EHCC Better When Combined DWI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University, China (Other)
Collaborators: First Hospital of China Medical University (Other)
Responsible Party: Principal Investigator, Xiaoping Yang, Principal Investigator, China Medical University, China
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: XYang
Record Dates: First submitted 2012-05-08; First posted 2012-05-09 (Estimated); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: Biliary Tract Neoplasm; Cholangiocarcinoma
Keywords: Biliary Tract Neoplasm; Cholangiocarcinoma; Diffusion magnetic resonance imaging; Magnetic resonance imaging; Magnetic resonance Cholangiopancreatography
MeSH Terms: conditions — Biliary Tract Neoplasms; Cholangiocarcinoma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Two experienced professors of radiology observed and analyzed the images separately. They were not involved in image acquisition and were blinded to the patients' clinical, surgical and histological information. Conventional MR sequences were qualitatively analyzed in the first reading session, including T2WI, FIESTA, 2D MRCP and 3D MRCP sequences, and after one week, DWI under three different b values with ADC map combined with the preceding conventional sequences were analyzed respectively as the second reading session.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- MRCP and DWI using 3T MRI (Experimental): MRCP and DWI using Magnetic resonance imaging（GE Signa,3.0 T )
  Interventions: Device: 3T MRI
- MRCP only using 3T MRI (Experimental): MRCP only using Magnetic resonance imaging（GE Signa,3.0 T )
  Interventions: Device: 3T MRI

INTERVENTIONS:
Device: 3T MRI — diffusion weighted imaging(DWI) of biliary tract with GE Signa 3-tesla device

SUMMARY:
Researching the diagnostic significance of Biliary Tract Neoplasm under combining DWI sequence with MRCP versus MRCP only separately.

DETAILED DESCRIPTION:
The purpose of the study is to evaluate the usefulness of diffusion weighted imaging(DWI) combined with MRCP of 3.0T magnetic resonance imaging (MRI) in the evaluation of suspected malignant bile duct diseases. People with suspected Biliary Tract Neoplasm based on clinical symptoms (such as jaundice and thinness with unknown reasons) and CA-199 value raises are included.Diagnosis divided into two steps: the first one，only provide conventional MR sequences and MRCP images to make a diagnosis; the second step,provide the DWI images additionally, combining the image data before to make a diagnosis. Hypothesis is that DWI sequence should be regularly added into MRCP examination for improving diagnosis rate of Biliary Tract Neoplasm.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Suspected Biliary Tract Neoplasm based on clinical symptoms(such as jaundice and thinness with unknown reasons)and CA-199 raises（>37U/mL）
* No evidence of clinical symptoms or CA-199 increase by non-bile duct cancerous factors(hepatitis,cholangeitis,stones)
* Age ≥ 16

Exclusion Criteria:

* Previous Biliary Tract Neoplasm surgery
* Contraindication for MRI (such as pacemaker or inner ear implant)
* Claustrophobia
* Age < 16

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2012-03 (Actual); Primary Completion 2013-03 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
EHCC performance on DWI, ADC map and MRCP | at the end of the study
  Two experienced professors of radiology observed and analyzed the images separately. If there were discrepancies, the two professors came to an agreement by consensus.

SECONDARY OUTCOMES:
ADC, SNR, CNR and SIR for EHCC lesion under different b values | at the end of the study
  The ADC value of EHCC in DWI under various b values was measured, and the SNR, the CNR and the SIR in DWI were calculated. The formula for calculating the ADC value was: ADC = [ln (S1 /S2)]/ (b2 -b1) , (S and b represent signal intensity and b value, 1 and 2 represent low and high, respectively).

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoping yang, MD, Principal Investigator — First Affiliated Hospital of China Medical University
Locations (1):
- Room of 3.0TMR in the FAH of CMU, Shenyang, Liaoning, China

IPD SHARING:
Plan to Share IPD: No